CLINICAL TRIAL: NCT02618239
Title: Effect of Prebiotics on Intestinal Gas Production, Microbiota and Digestive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PR(AG)296/2013
Record Dates: First submitted 2015-11-11; First posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: intestinal gas; Healthy subjects; microbiota; prebiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy subjects (Experimental): Bimuno Galacto-oligo-saccharide administration 2.7 g/d x 3 weeks
  Interventions: Dietary Supplement: Bimuno Galacto-oligo-saccharide

INTERVENTIONS:
Dietary Supplement: Bimuno Galacto-oligo-saccharide

SUMMARY:
Non-absorbable, fermentable residues in the diet increase intestinal gas production and induce gas-related symptoms, such as flatulence, abdominal bloating and distention; however, prebiotics, which are also fermented by colonic bacteria have been shown to improve this type of symptoms. The aim is to demonstrate changes in metabolic activity of gut microbiota and colonic biomass induced by prebiotics.

Healthy subjects (n=20) will be administered a prebiotic (Galacto-oligo-saccharide; 2.8 g/d) for 3 weeks; they will also receive a standard diet during three days. The following outcomes will be measured immediately before, at the beginning and at the end of the treatment: a) number of gas evacuations during daytime for 2 days on the standard diet, by means of an event marker; b) volume of gas evacuated via a rectal tube during 4 hours after a test meal, by means of a barostat; c) microbiota composition by fecal analysis.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* gastrointestinal symptoms
* recent (3 months) antibiotic intake
* recent (3 months) change of diet
* recent (3 months) gastroenteritis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of daily anal gas evacuations | Change from beginning of treatment (mean of days 2 and 3) to end of treatment (mean of days 20 and 21)

SECONDARY OUTCOMES:
Volume of anal gas evacuation | Change from beginning of treatment (day 3) to end of treatment (day 21)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Azpiroz, MD, Principal Investigator — Vall d'Hebron Research Institute

REFERENCES:
- [Derived] Mego M, Manichanh C, Accarino A, Campos D, Pozuelo M, Varela E, Vulevic J, Tzortzis G, Gibson G, Guarner F, Azpiroz F. Metabolic adaptation of colonic microbiota to galactooligosaccharides: a proof-of-concept-study. Aliment Pharmacol Ther. 2017 Mar;45(5):670-680. doi: 10.1111/apt.13931. Epub 2017 Jan 12. PMID 28078750